CLINICAL TRIAL: NCT00503815
Title: A Safety and Efficacy Evaluation of BLI-800 vs an Active Control Bowel Preparation in Adult Subjects Undergoing Colonoscopy
Brief Title: BLI-800-302: BLI-800 vs an Active Control Bowel Preparation in Adult Subjects Undergoing Colonoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Responsible Party: John McGowan, Clinical Operations Manager, Braintree Laboratories, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: BLI-800-302
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Last update posted 2007-12-27 (Estimated); Status verified 2007-12

CONDITIONS: Colonoscopy
Keywords: colonoscopy; bowel preparation; prep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: BLI-800
Drug: Polyethylene glycol 3350 based bowel preparation

SUMMARY:
This is a randomized, parallel, multi-center, single-blind study, comparing BLI-800 to an FDA approved bowel preparation in adult subjects undergoing colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

-Male or female outpatients who are undergoing colonoscopy for a routinely accepted indication, including:

Evaluation of BE results GI bleeding Anemia of unknown etiology Neoplastic disease surveillance Endosonography Inflammatory bowel disease Unknown diarrhea or constipation etiology Polypectomy Laser therapy Routine Screening

* At least 18 years of age
* Otherwise in good health, as determined by physical exam and medical history
* If female, and of child-bearing potential, is using an acceptable form of birth control (hormonal birth control, IUD, double-barrier method, depot contraceptive, abstinent, or vasectomized spouse)
* Negative urine pregnancy test at screening, if applicable
* In the Investigator's judgment, subject is mentally competent to provide informed consent to participate in the study

Exclusion Criteria:

* Subjects with known or suspected ileus, severe ulcerative colitis, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis, or megacolon.
* Subjects with impaired consciousness that predisposes them to pulmonary aspiration.
* Subjects who are undergoing colonoscopy for foreign body removal and decompression.
* Subjects with clinically significant electrolyte abnormalities based on Visit 1 laboratory results, such as hypernatremia, hyponatremia, hyperphosphatemia, hypokalemia, hypocalcemia, dehydration, or those secondary to the use of diuretics or angiotensin converting enzyme (ACE) inhibitors.
* Subjects with a history of renal or hepatic insufficiency or congestive heart failure.
* Subjects who had previous gastrointestinal surgeries
* Subjects who are pregnant or lactating, or intending to become pregnant during the study.
* Subjects of childbearing potential who refuse a pregnancy test.
* Subjects who are allergic to any preparation components
* Subjects who, in the opinion of the Investigator, should not be included in the study for any reason, including inability to follow study procedures.
* Subjects who have participated in an investigational clinical, surgical, drug, or device study within the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2007-07; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Efficacy - preparation quality using a 4 point scale | 2-Day

SECONDARY OUTCOMES:
Safety-preparation related side effects; laboratory analysis | 30-Day

CONTACTS AND LOCATIONS:
Overall Officials: John D McGowan, B.S., Study Director — Braintree Laboratories, Inc.
Locations (10):
- United States (10):
  - Anaheim, California
  - Orange, California
  - Jackson, Mississippi
  - Portland, Oregon
  - Franklin, Tennessee
  - Germantown, Tennessee
  - Jackson, Tennessee
  - Nashville, Tennessee
  - Houston, Texas
  - Bellevue, Washington